CLINICAL TRIAL: NCT02171013
Title: Bioequivalence of Two Different Drug Product Batches of 150 mg of Dabigatran Etexilate Following Oral Administration in Healthy Male and Female Volunteers (Double Blind, Randomised, Single-dose, Replicate Design in a Two-treatments, Four Periods Crossover Study)
Brief Title: Bioequivalence of Two Different Drug Product Batches of Dabigatran Etexilate Following Oral Administration in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.56
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- Dabigatran etexilate batch A (Experimental)
  Interventions: Drug: Dabigatran polymorph I (≈ 83%) and polymorph II (≈17%)
- Dabigatran etexilate batch B (Experimental)
  Interventions: Drug: Dabigatran polymorph I

INTERVENTIONS:
Drug: Dabigatran polymorph I (≈ 83%) and polymorph II (≈17%)
  Arms: Dabigatran etexilate batch A
Drug: Dabigatran polymorph I
  Arms: Dabigatran etexilate batch B

SUMMARY:
To establish the bioequivalence of two drug product batches of dabigatran etexilate, one batch containing only polymorph I vs. the other batch containing 17% of dabigatran etexilate polymorph II in addition to polymorph I

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥65 and ≤85 years
3. BMI ≥18.5 and BMI ≤32.0 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Clinically relevant surgery of gastrointestinal tract
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. Any relevant bleeding history
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within four weeks prior to administration or during the trial
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Inability to comply with dietary regimen of study centre

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of total BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 72 hours after drug administration
Maximum measured concentration of total BIBR 953 ZW in plasma (Cmax) | Up to 72 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of free BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 72 hours after drug administration
Maximum measured concentration of free BIBR 953 ZW in plasma (Cmax) | Up to 72 hours after drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | Up to 72 hours after drug administration
Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2 (AUCt1-t2) | t1 = 0 and t2 = 24, 48, 72 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | Up to 72 hours after drug administration
Terminal rate constant in plasma (λz) | Up to 72 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 72 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | Up to 72 hours after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F ) | Up to 72 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | Up to 72 hours after drug administration
Change from baseline in physical examination | Baseline, day 73
Change from baseline in vital signs (blood pressure, pulse rate) | Baseline, day 73
Change from baseline in 12-lead ECG (electrocardiogram) | Baseline, day 73
Change from baseline in clinical laboratory tests | Baseline, day 73
Number of Participants with Serious and Non-Serious Adverse Events | Up to day 73
Assessment of tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Day 73